CLINICAL TRIAL: NCT02985294
Title: DOLORisk: Understanding Risk Factors and Determinants for Neuropathic Pain - Peripheral Physiological Measures as Determinants of Pain Risk
Brief Title: Peripheral Physiological Measures as Determinants of Pain Risk
Acronym: DOLORiskWP51
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neuroscience Technologies SLP, Barcelona (Industry)
Collaborators: University of Oxford (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Aarhus (Other); University of Dundee (Other)
Responsible Party: Sponsor
Other Study IDs: Neuroscience Technologies
Record Dates: First submitted 2016-11-28; First posted 2016-12-07 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Polyneuropathies; Peripheral Nerve Injuries; Peripheral Nervous System Diseases; Chemotherapy Effects; Neuralgia
Keywords: Neuropathic pain; Quantitative Sensory Testing; Multiple Excitability Measures; Threshold Tracking
MeSH Terms: conditions — Polyneuropathies; Peripheral Nerve Injuries; Peripheral Nervous System Diseases; Neuralgia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — blood sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cross-sectional cohort: Multiple Excitability Measures of peripheral nerves on patients with chronic peripheral neuropathic pain
  Interventions: Other: Multiple Excitability Measures of peripheral nerves
- Longitudinal cohort: Multiple Excitability Measures of peripheral nerves on painless patients before and after potential chronic neuropathic pain-inducing interventions (chemotherapy, surgery)
  Interventions: Other: Multiple Excitability Measures of peripheral nerves

INTERVENTIONS:
Other: Multiple Excitability Measures of peripheral nerves — The technique of threshold tracking can be used to obtain several measures of peripheral nerve excitability (Multiple Excitability Measures or MEM), such as refractoriness, supernormality, strength-duration time constant and 'threshold electrotonus' (i.e. the changes in threshold produced by long-lasting depolarizing or hyperpolarizing current pulses). Each of these measurements depends on membrane potential and on other biophysical properties of the axons. Many of these excitability parameters are very constant among different subjects, while other, such as the current/threshold parameters and the super/sub-excitability parameters, appear to be characteristic of an individual
  Other Names: Assessment of sensory phenotype by QST (quantitative sensory testing); Questionnaires

SUMMARY:
This study evaluates peripheral nervous system function using Multiple Excitability Measures (MEM) to obtain "electrophysiological pain phenotypes"

DETAILED DESCRIPTION:
Using MEM for peripheral sensory and motor axons we want to identify a set of excitability measures that:

1. Correlate with parameters of clinical pain and of pain processing in existing pain patients (cross sectional study), with the aim to obtain an objective Pain Biomarker.
2. Predict development of neuropathic pain in susceptible patients (longitudinal study). Neuropathic Pain Predictor for patients:

i. Undergoing surgical procedures associated with a relatively high risk of developing neuropathic pain such as thoracotomy and hernia repair ii. Planning to start chemotherapy with potentially neurotoxic agents such as vincristine

ELIGIBILITY:
Inclusion Criteria:

* Chronic peripheral neuropathic pain
* Painless Patient with risk to develop neuropathic pain (post-surgery, chemotherapy-induced)

Exclusion Criteria:

* Minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Painless patients and patients with chronic peripheral neuropathic pain
  2. Susceptible patients for developing pain i. Undergoing surgical procedures associated with a relatively high risk of developing neuropathic pain such as thoracotomy and hernia repair ii. Planning to start chemotherapy with potentially neurotoxic agents such as taxol, vincristine, etc.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-03 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Electrophysiological pain phenotypes using MEM. Pain biomarker | Single assessment (cross sectional study) at the first and only visit
  Correlate with parameters of clinical pain and of pain processing in existing pain patients
Electrophysiological pain phenotypes using MEM. Pain predictor | Single assessment at baseline, before any procedure (surgery/chemotherapy)
  Predict development of neuropathic pain in susceptible patients

CONTACTS AND LOCATIONS:
Locations (1):
- Neuroscience technologies, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No